CLINICAL TRIAL: NCT04968990
Title: Multi-Center Trial Sponsored by St. Jude Children's Research Hospital for the Treatment of Newly Diagnosed Patient's With Wilm's Tumor Requiring Abdominal Radiation Delivered With Proton Beam Irradiation
Brief Title: Treatment of Newly Diagnosed Patient's With Wilm's Tumor Requiring Abdominal Radiation Delivered With Proton Beam Irradiation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJWT21
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Wilms Tumor
Keywords: Retroperitoneum; Retroperitoneal subsites; Kidney; Lymph node involvement; Abdomen
MeSH Terms: conditions — Wilms Tumor | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Favorable Histology Stage I & II and FH Stage III/IV (Active Comparator): Favorable Histology Stage I & II and FH Stage III/IV Delayed Local Control with clear surgical margins and pathologically negative lymph nodes. Participants will undergo complete surgical resection at diagnosis or after 6-12 weeks of induction chemotherapy.
  Interventions: Procedure: Complete Surgical Resection
- Stage III & IV Adjuvant RT and Stage V (Active Comparator): Participants will undergo surgical resection at diagnosis or after 6-12 weeks of induction chemotherapy. Those with evidence of LN involvement, surgical margin involvement, local or diffuse spill, gross disease in the renal bed or peritoneal implants, will receive adjuvant PBRT.
  Interventions: Device: Proton Beam Radiation (PBRT); Drug: DD-4A Chemotherapy Regimen; Procedure: Surgical Resection
- Stage V Adjuvant RT: (Active Comparator): Participants will undergo partial nephrectomy after 6-12 weeks of induction chemotherapy. Those with evidence of LN involvement, surgical margin involvement, local or diffuse spill, gross disease in the renal bed or peritoneal implants, will receive adjuvant PBRT
  Interventions: Device: Proton Beam Radiation (PBRT); Drug: DD-4A Chemotherapy Regimen; Procedure: Partial Nephrectomy

INTERVENTIONS:
Device: Proton Beam Radiation (PBRT) — The treatment approach with radiation therapy prescribed in this trial is designed to deliver highly conformal radiation therapy (proton beam radiation or intensity modulated photon radiation) to target volumes that are based on the burden of disease.
  Arms: Stage III & IV Adjuvant RT and Stage V; Stage V Adjuvant RT:
Drug: DD-4A Chemotherapy Regimen — Patients will receive standard of care chemotherapy based on diagnosis and stage.
  Arms: Stage III & IV Adjuvant RT and Stage V; Stage V Adjuvant RT:
Procedure: Complete Surgical Resection — Participants will undergo complete surgical resection at diagnosis or after 6-12 weeks of induction chemotherapy
  Arms: Favorable Histology Stage I & II and FH Stage III/IV
Procedure: Surgical Resection — Participants will undergo surgical resection at diagnosis or after 6-12 weeks of induction chemotherapy.
  Arms: Stage III & IV Adjuvant RT and Stage V
Procedure: Partial Nephrectomy — Participants will undergo partial nephrectomy after 6-12 weeks of induction chemotherapy.
  Arms: Stage V Adjuvant RT:

SUMMARY:
Participants are being asked to take part in this clinical trial, a type of research study, because the participants have a Wilms Tumor cancer.

Primary Objectives

To determine whether delivery of proton beam radiation to a conformal reduced target volume in the flank allows normal flank growth compared to the contralateral untreated side and non-irradiated patients.

Secondary Objectives

To deliver proton beam radiation to a conformal reduced target volume (partial kidney proton beam radiation therapy) in the affected kidney(s) for patients with Stage V (bilateral Wilms tumor) and specific involved surgical margins yielding no reduction in the high control rates seen with more traditional flank / whole kidney fields.

Exploratory Objectives

* Study the feasibility of sparing the residual kidney, spine and liver in patients requiring whole abdomen radiation therapy using either a proton beam treatment technique or intensity-modulated radiation therapy ( IMRT) photon based technique.
* Study the feasibility of delivering whole lung radiation therapy with proton beams with the goals of sparing the developing breast tissue, heart structures, thyroid and liver.
* Develop simultaneous xenografts and organoid models from the same starting material to study Wilms tumor biology and compare responses to chemotherapeutic agents.
* Define the evolution of organ specific (kidney, liver, pancreas, etc.) abnormalities (laboratory studies) as an early marker of possible late end organ damage and their relationship to radiation.
* Study and evaluate impact of proton therapy on the musculoskeletal system and physical performance and compare with photon therapy cases treated with classical treatment fields.
* Assess CTC-AE and Pediatric Patient Reported Outcomes during radiation and in follow-up, correlating with disease, treatment and patient variables.
* Correlate quantitative MRI values, including apparent diffusion coefficient (ADC) values, with histopathology findings post-surgery in children with (bilateral) Wilms.
* Assess daily variations in proton range along each treatment beam using standard pre-treatment cone beam CT or on-treatment MR.

DETAILED DESCRIPTION:
Participants will receive proton beam radiation therapy (PBRT) according to stage and surgical findings.

Favorable Histology Stage I & II and FH Stage III/IV Delayed Local Control with clear surgical margins and pathologically negative lymph nodes: Participants will undergo complete surgical resection at diagnosis or after 6-12 weeks of induction chemotherapy. PBRT will not be administered to the primary site in those with no evidence of spill, peritoneal involvement, lymph node (LN) involvement or microscopic residual in the abdomen. Systemic therapy will be delivered in a standard of care manner according to histology and stage.

Stage III & IV Adjuvant RT: Participants will undergo surgical resection at diagnosis or after 6-12 weeks of induction chemotherapy. Those with evidence of LN involvement, surgical margin involvement, local or diffuse spill, gross disease in the renal bed or peritoneal implants, will receive adjuvant PBRT. Systemic therapy will be delivered in a standard of care manner according to histology and stage.

Stage V Adjuvant RT: Participants will undergo partial nephrectomy after 6-12 weeks of induction chemotherapy. Those with evidence of LN involvement, surgical margin involvement, local or diffuse spill, gross disease in the renal bed or peritoneal implants, will receive adjuvant PBRT. Systemic therapy will be delivered in a standard of care manner according to histology and stage.

Systemic therapy will follow a well-defined standard of care based on Children's Oncology Group (COG) approaches including pre-operative chemotherapy and adjuvant chemotherapy. The intent will be to standardize chemotherapy to ensure a consistent background of standard of care therapy, while not mandating additional data collection beyond the specific trial objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible to be enrolled on this trial at the time of initial (or presumptive) diagnosis of Wilms tumor, at the time of surgery or at the time of radiation treatment.
* Patients that are determined to be stage I or II will be eligible for the surgical and biologic aspects of this trial but will otherwise be followed per institutional standards and be "off therapy" at the time of stage determination (followed only for survival).
* Patients identified to have an anaplastic or other unfavorable tissue component (non-Wilms histology) to their tumor may have tissue assessed for the biology objective but will be removed from the therapeutic portion of the study at the time of identification of this pathologic finding.

Performance Level • The Karnofsky performance status must be ≥50 for patients >16 years of age and the Lansky performance status must be ≥ 50 for patients ≤ 16 years of age.

Prior Therapy

* Only prior therapy with the initial chemotherapy regimen defined in section 5.1 and Appendix III are allowed for patients that are treated with neoadjuvant chemotherapy. These patients may change to an alternate regime based on response or biologic features and noted in section 5.1. Prior biopsy or surgery is allowed.
* Prior radiation therapy is not allowed if directed at the abdomen. Emergent RT to other sites of disease is acceptable.

Organ Function Requirements:

* None - As per institutional standard of care. Diagnosis / Stage
* Presumed diagnosis of Wilms tumor (continued management on trial will depend on stage and histology)
* Resected upfront stage III, IV or V favorable histology Wilms tumor. Stage III includes any one or multiples of the following:

  * Lymph nodes within the abdomen or pelvis are involved by tumor. (Lymph node involvement in the thorax, or other extra-abdominal sites is a criterion for Stage IV)
  * The tumor has penetrated through the peritoneal surface
  * Tumor implants are found on the peritoneal surface
  * Gross or microscopic tumor remains post-operatively (e.g., tumor cells are found at the margin of surgical resection on microscopic examination - in the post chemotherapy setting only specific types of viable tumor at the surgical margin are considered stage III AND require adjuvant radiation - see surgery / pathology / radiation section for additional details)
  * The tumor is not completely resectable because of local infiltration into vital structures
  * Tumor spillage occurring either before or during surgery
  * A trans abdominal biopsy (regardless of type- tru-cut, open or fine needle aspiration) was performed prior to resection or chemotherapy. Retroperitoneal biopsies DO NOT require radiotherapeutic management like stage III
  * Tumor is removed in greater than one piece (e.g. tumor cells are found in a separately excised adrenal gland; a tumor thrombus within the renal vein is removed separately from the nephrectomy specimen). Extension of the primary tumor within vena cava into thoracic vena cava and heart is considered Stage III, rather than Stage IV even though outside the abdomen.
* Stage IV - Hematogenous metastases (lung, liver, bone, brain, etc.), or lymph node metastases outside the abdomino-pelvic region are present. (The presence of tumor within the adrenal gland is not interpreted as metastasis and staging depends on all other staging parameters present). Patients with lung involvement and local abdominal stage I or II are eligible to remain on trial for whole lung irradiation objective.
* Stage V - Bilateral renal involvement by tumor is present at diagnosis. An attempt should be made to stage each side according to the above criteria on the basis of the extent of disease
* Patients that have or will receive neoadjuvant chemotherapy for unresected unilateral or bilateral Wilms tumor without a biopsy are not assumed to be require adjuvant radiation on this study. That determination will be based on surgical findings and the approach to treatment detailed in the protocol.

Timing

* Patients undergoing upfront surgery must start RT, if indicated, within 28 days of definitive surgery with a goal of starting RT by day 21.
* Patients receiving neoadjuvant chemotherapy will be enrolled either at diagnosis (if at St. Jude) or at the time of RT.

Other Criteria

• Female patients of childbearing potential (age ≥10 years old or post-menarche) must have a negative pregnancy test prior to enrollment.

Exclusion Criteria:

* Inability or unwillingness to provide written informed consent
* Prior radiation therapy to a site to be treated with proton / photon radiation as part of this trial. Emergent radiation is allowed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Half circumference at 3 year | 3 years after all patients finish proton therapy
  Half circumference measurement at 3 year from irradiated and unirradiated hemi-abdomen for patients in need of flank radiation
Half circumference at 5 year | 5 years after all patients finish proton therapy
  Half circumference measurement at 5 year from irradiated and unirradiated hemi-abdomen for patients in need of flank radiation
Half circumference at 7 year | 7 years after all patients finish proton therapy
  Half circumference measurement at 7 year from irradiated and unirradiated hemi-abdomen for patients in need of flank radiation
Half circumference at 10 year | Half circumference measurement at 10 year from irradiated and unirradiated hemi-abdomen
  Half circumference measurement at 10 year from irradiated and unirradiated hemi-abdomen for patients in need of flank radiation

SECONDARY OUTCOMES:
Local control rate in a partially radiated kidney | 5 years
  This objective is to investigate whether deliver proton beam radiation to a conformal reduced target volume (partial kidney proton beam radiation therapy) in the affected kidney(s) for patients Stage V (bilateral Wilms tumor) with specific involved surgical margins yielding no reduction in the high control rates seen with more traditional flank / whole kidney fields.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Krasin, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St.Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St.Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols